CLINICAL TRIAL: NCT02708667
Title: An Observational Research on Relationship Between c-Met Gene Polymorphism, Promoter Methylation Level, Related Drug Metabolism Enzymes and Crizotinib's Hepatic Toxicity in Non-small Cell Lung Cancer Patients
Brief Title: An Observational Research Of Crizotinib's Hepatic Toxicity In Non-small Cell Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Associate Professor/Associate chief physician, Sun Yat-sen University
Other Study IDs: 2015-FXY-078-Internal medicine
Record Dates: First submitted 2016-03-05; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; crizotinib; hepatic toxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood, biopsy tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Crizotinib, an inhibitor of anaplastic lymphoma kinase (ALK), was approved by Food and Drug Administration (FDA) for the treatment of patients with ALK-positive non-small cell lung cancer (NSCLC) and its administration has achieved considerable success. However, adverse effects inevitably occurred and the most common one was hepatic toxicity, appearing as elevating alanine aminotransferase(ALT) and aspartate aminotransferase(AST). Therefore, the investigators try to figure out the mechanism of crizotinib-inducing hepatic toxicity, and explore whether there is any biological marker to diagnose this side effect in an early stage, which may realize individualized therapy with more efficacy and less side effects.

ELIGIBILITY:
Inclusion Criteria:

1. patients who were histologically and cytologically confirmed NSCLC at stage III or IV
2. harbored ALK fusion gene and took crizotinib
3. age:18~75years
4. Eastern cooperative oncology group performance status(ECOG PS): 0~2 points
5. the expected lifetime is more than 12 weeks after being recruited

Exclusion Criteria:

1. patients who also suffered from other malignant tumor
2. uncontrolled systemic diseases,central nervous system (CNS) metastasis
3. clinically active interstitial lung diseases
4. severe liver dysfunction caused by hepatic cirrhosis or hepatitis （Child-Pugh class C, total index score 10-15 points）
5. taking drugs that interact with crizotinib

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with stage III or IV non-small cell lung cancer (NSCLC), harbored ALK fusion gene and took crizotinib.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
number of patients with adverse events | change from the date of taking crizotinib at 9 months

SECONDARY OUTCOMES:
progression free survival | from the date of taking crizotinib to the date of objective tumor progression or date of death from any cause,whichever came first,assessed up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Likun Chen, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China